CLINICAL TRIAL: NCT04026334
Title: Evaluation of Hydromechanical Cleansing Using Normal Saline With V.A.C. VERAFLO CLEANSE CHOICE™ Dressing and NPWT-d to Promote Increased Healthy Wound Bed Tissue
Brief Title: Evaluation of V.A.C. VERAFLO CLEANSE CHOICE™ Dressing Using Normal Saline to Promote Increased Healthy Wound Bed Tissue
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient subject accrual rate
Sponsor: 3M (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCI.CLEANSE.CHOICE.2019.01
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Wound; Wound Heal; Wounds and Injuries; Granulation Tissue; Negative-pressure Wound Therapy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- V.A.C. VERAFLO CLEANSE CHOICE™ with Normal Saline (Experimental)
  Interventions: Device: V.A.C. VERAFLO CLEANSE CHOICE™ dressing with Normal Saline

INTERVENTIONS:
Device: V.A.C. VERAFLO CLEANSE CHOICE™ dressing with Normal Saline — -125mmHg, 10 minute soak time, 3.5 hours of negative pressure therapy

SUMMARY:
The study goal is to evaluate the ability of the V.A.C. ULTA™ Negative Pressure Wound Therapy System and V.A.C. VERAFLO CLEANSE CHOICE ™ (VFCC) dressing system with saline as an irrigant in increasing viable tissue in full thickness wounds (such as chronic, acute, traumatic, sub-acute, and dehisced wounds and/or ulcers) with difficult to manage bioburden and slough.

ELIGIBILITY:
Inclusion Criteria:

1. is anticipated to be hospitalized for the duration of treatment.
2. is ≥22 years of age or their legally authorized representative is able to provide informed consent.
3. has a full thickness wound (such as chronic, acute, traumatic, sub-acute, and dehisced wounds and/or ulcers) measuring ≥4cm in length and ≥4cm in width (before removal of eschar at the bedside) excluding undermining/tunneling.
4. has, in the opinion of the investigator, no more than 2/3 of the visible wound bed surface area considered to be clean, healthy, and viable. If eschar is present at baseline, it must be removed by bedside debridement prior to assessing the percentage of clean, healthy, and viable wound bed.
5. has a negative urine or serum pregnancy test at screening (if female and has potential for pregnancy) and is willing to take precautionary measures to prevent pregnancy during the duration of the study (up to 9 days).

Exclusion Criteria:

1. has been diagnosed with malignancy in the wound.
2. has untreated osteomyelitis.
3. has an untreated systemic infection.
4. has active cellulitis in the peri wound area.
5. has a known allergy or hypersensitivity to study materials: dressing and/or dressing components such as acrylic adhesives or polyurethane.
6. has, in the opinion of the investigator, a clinically significant condition that would impair the Subject's ability to comply with the study procedures.
7. has had radiation directly to the wound.
8. has been diagnosed with a major vascular deficit limiting arterial inflow to the wound region, as determined by the Investigator's interpretation of the Subject's medical history.
9. has eschar in the wound that cannot be removed by beside or sharp and/or mechanical debridement.
10. is participating in another interventional clinical trial for the duration of the study.
11. has unexplored fistulas in the wound or fistulas in the wound that connect to other body cavities.
12. has inadequate hemostasis at the wound site, as determined by the investigator.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Percent change in wound bed surface area (cm2) of clean, healthy, viable tissue | Baseline to Day 6-9

SECONDARY OUTCOMES:
Percent change in total wound volume (cm3) | Baseline to Day 6-9
Percent change in total wound area (cm2) | Baseline to Day 6-9
Physician assessment of the need for surgical debridement | Day 6-9
  This will be a subjective assessment made by the Investigator of Yes or No

CONTACTS AND LOCATIONS:
Locations (1):
- Joseph M. Still Research Foundation, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No